CLINICAL TRIAL: NCT06641986
Title: Identification and Validation of a Prediction Model of Postoperative Anxiety Symptom in Elderly Patients Undergoing Major Noncardiac Surgery: a Prospective Multicenter Cohort Study
Brief Title: A Prediction Model of Postoperative Anxiety Symptom in Elderly Patients Undergoing Major Noncardiac Surgery
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Peking University First Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Xiangya Hospital of Central South University (Other); Beijing Anzhen Hospital (Other); Central South University (Other); Peking University People's Hospital (Other); Zhejiang University (Other); Fudan University (Other); Sun Yat-sen University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); China-Japan Friendship Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Taihe Hospital (Other); Zhejiang Provincial People's Hospital (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-AN-001
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-08

CONDITIONS: Predictive Model
Keywords: predicted model; major non-cardiac surgery; elderly patients; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly patients: elderly patients undergoing major non-cardiac surgery (aged ≥ 65 years)

SUMMARY:
A multicentre, prospective observational study to develop and validate a predictive model for postoperative anxiety symptoms in elderly Chinese patients undergoing non-cardiac major surgery.

DETAILED DESCRIPTION:
In 2015, the WHO introduced the concept of "healthy ageing" for global ageing, with a focus on the mental health of older people at its core. More than 20 million elderly patients undergo surgery each year in China, accounting for a quarter of the population who undergo surgery. Previous studies have found high risk of anxiety in older perioperative patients, especially for non-cardiac major surgery patients. Therefore, it is necessary to construct a predictive model of anxiety in elderly patients undergoing non-cardiac major surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients (age ≥ 65 years).
2. Undergoing elective surgery with a planned overnight hospital stay following surgery.
3. Major non-cardiac surgery, non-neurosurgical surgery.

Exclusion Criteria:

1. History of previous severe mental illness or long-term use of psychotropic medications.
2. Immediately admitted to ICU after surgery.
3. Death within 7 days after surgery.
4. Grade of surgery ≤ 2.
5. Failure to complete the postoperative anxiety assessment.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients (aged ≥ 65 years) who completed the anxiety and depression assessment after the elective major noncardiac, non-neurosurgical surgery were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 5551 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Anxiety | within 7 days after surgery
  The GAD-7 is a seven-item questionnaire for screening on the presence of generalized anxiety disorder and assessing its severity. Items were scored on a four-point scale with total scores ranging from zero to twenty-one. Scores were defined as: ≥5 mild, ≥10 moderate, and ≥15 severe anxiety. The recommended screening cutoff was ≥10, corresponding with at least a moderate level of anxiety. Higher scores mean more anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- First Medical center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided